CLINICAL TRIAL: NCT05085314
Title: Prospective Multicenter Randomized Controlled 1:1 Study Evaluating the Efficacy of a 3D Digital Operating Microscope Compared to Conventional Microscopes Microscopes on the Comfort and Subjective Visual Sensations of the Patients Related to the Microscope Light During Initial Cataract Surgery Under Topical Anesthesia Topical Anesthesia
Brief Title: Comfort Operative Ocular Light Study
Acronym: COOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTI_2021_7
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cataract
Keywords: Ngenuity 3D digital operating system
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ngenuity digital 3D microscope (Experimental)
  Interventions: Procedure: Ngenuity digital 3D microscope
- Conventional microscope (Active Comparator)
  Interventions: Procedure: Conventional microscope

INTERVENTIONS:
Procedure: Ngenuity digital 3D microscope — Cataract surgery under topical anesthesia with the Ngenuity digital 3D microscope, Alcon, Fort Worth, TX
  Arms: Ngenuity digital 3D microscope
Procedure: Conventional microscope — Cataract surgery under topical anesthesia with a conventional microscope
  Arms: Conventional microscope

SUMMARY:
Digital 3D microscopes require less light and may be more comfortable for patients requiring cataract surgery under topical anesthesia compared to conventional microscopes.

To date, no studies have evaluated the comfort and subjective visual sensations related to the light of the 3D digital microscope in cataract surgery patients.

The purpose of this study is to evaluate the effectiveness of the Ngenuity 3D digital operating system (Alcon, Fort Worth, TX) compared to conventional microscopes on the comfort and subjective visual sensations related to of patients undergoing initial cataract surgery under topical anesthesia (pure or combined with intravenous sedation).

DETAILED DESCRIPTION:
Patients will be recruited during the preoperative consultation where the indication for cataract surgery. The allocation of the management arm (3D digital microscope or conventional microscope) will be randomized in a stratified way on the center.

Prior to his or her operative session, the surgeon will set up the microscope with his or her usual parameters.

The light intensity will be measured at the beginning of the operating session with a calibrated light meter. The type of anesthesia (pure topical or associated with intravenous sedation), the duration of the operation, intraoperative complications (frequency and type), and the possible use of an anesthesiologist to inject additional intravenous anesthetic will be collected.

Before the patient is discharged from the ambulatory surgical unit, the clinical study technician will ask the patient the 4 questions of the standardized questionnaire assessing comfort and subjective visual sensations related to the microscope light.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a first surgery (= first eye to be operated) of cataract alone under topical anesthesia (pure or associated with intravenous sedation)
* Express consent to participate in the study

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Patient with comprehension problems or who does not understand French well
* Pregnant or breastfeeding woman
* Indication for another surgery on the operated side (e.g. vitrectomy combined with cataract surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Glare of patients related to the light of the microscope of the patients | two hours maximum after surgery
  Patient response to the question "Were you dazzled by light during surgery?" rated on a numerical scale from 0 (Not at all) to 10 (Yes, very much)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin TADAYONI, Principal Investigator — Hôpital Fondation A. de Rothschild; Vincent GUALINO, Study Chair — Clinique Honoré Cave, Montauban; Aude COUTURIER, Study Chair — Hôpital Lariboisière
Locations (2):
- France (2):
  - Clinique Honoré Cave, Montauban
  - Hôpital Fondation A. de Rothschuld, Paris

REFERENCES:
- [Derived] Gualino V, Pierne K, Manassero A, Bruneau S, Couturier A, Tadayoni R. Comparing microscope light-associated glare and comfort between heads-up 3D digital and conventional microscopes in cataract surgery: a randomised, multicentre, single-blind, controlled trial. BMJ Open Ophthalmol. 2023 Jun;8(1):e001272. doi: 10.1136/bmjophth-2023-001272. Epub 2023 Jun 26. PMID 37493673